CLINICAL TRIAL: NCT01702571
Title: A Two-Cohort, Open-Label, Multicenter Study of Trastuzumab Emtansine (T-DM1) in HER2-Positive Locally Advanced or Metastatic Breast Cancer Patients Who Have Received Prior Anti-HER2 and Chemotherapy-Based Treatment
Brief Title: A Study of Trastuzumab Emtansine in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Breast Cancer Who Have Received Prior Anti-HER2 And Chemotherapy-based Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO28231; 2012-001628-37 (EudraCT Number)
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Results first posted 2021-08-05 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trastuzumab Emtansine (All Participants) (Experimental): This cohort will enroll all participants with HER2-positive, unresectable, LABC or mBC who have received prior anti-HER2 and chemotherapy treatment and have progressed on or after the most recent treatment for LABC or mBC, or within 6 months of completing adjuvant therapy. Participants will receive trastuzumab emtansine every 3 weeks until unacceptable toxicity, withdrawal of consent, or disease progression.
  Interventions: Drug: Trastuzumab Emtansine
- Trastuzumab Emtansine (Asian Participants) (Experimental): This cohort will enroll Asian race participants with HER2-positive, unresectable, LABC or mBC who have received prior anti-HER2 and chemotherapy treatment and have progressed on or after the most recent treatment for LABC or mBC, or within 6 months of completing adjuvant therapy. Participants will receive trastuzumab emtansine every 3 weeks until unacceptable toxicity, withdrawal of consent, or disease progression.
  Interventions: Drug: Trastuzumab Emtansine

INTERVENTIONS:
Drug: Trastuzumab Emtansine — Participants will receive trastuzumab emtansine 3.6 milligrams per kilogram (mg/kg) intravenously on Day 1 of a 3-week cycle every 3 weeks until unacceptable toxicity, withdrawal of consent, or disease progression.
  Other Names: RO5304020, T-DM1, Kadcyla

SUMMARY:
This two-cohort, open-label, multicenter study will assess the safety, efficacy and tolerability of trastuzumab emtansine in participants with HER2-positive locally advanced breast cancer (LABC) or metastatic breast cancer (mBC) who have received prior anti-HER2 and chemotherapy-based treatment. Participants in Cohort 1 will be drawn from the general participant population; Cohort 2 will include only Asian participants.

ELIGIBILITY:
Inclusion Criteria:

* HER2-positive disease determined locally
* Histologically or cytologically confirmed invasive breast cancer
* Prior treatment for breast cancer in the adjuvant, unresectable, locally advanced or metastatic setting must include both chemotherapy, alone or in combination with another agent, and an anti-HER2 agent, alone or in combination with another agent
* Documented progression of incurable, unresectable, LABC, or mBC, defined by the investigator: progression must occur during or after most recent treatment for LABC/mBC or within 6 months of completing adjuvant therapy
* Measurable and/or non-measurable disease
* Left ventricular ejection fraction (LVEF) >/=50% by either echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2
* Adequate organ function
* Use of highly effective contraception as defined by the protocol

Exclusion Criteria:

* History of treatment with trastuzumab emtansine
* Prior enrollment into a clinical study containing trastuzumab emtansine regardless of having received trastuzumab emtansine or not
* Peripheral neuropathy of Grade >/= 3 per National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) v 4.0
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage 1 uterine cancer, synchronous or previously diagnosed HER2-positive breast cancer
* History of receiving any anti-cancer drug/biologic or investigational treatment within 21 days prior to first study treatment except hormone therapy, which can be given up to 7 days prior to first study treatment; recovery of treatment-related toxicity consistent with other eligibility criteria
* History of exposure to cumulative doses of anthracyclines
* History of radiation therapy within 14 days of first study treatment. The participant must have recovered from any resulting acute toxicity (to Grade </=1) prior to first study treatment.
* Metastatic central nervous system (CNS) disease only
* Brain metastases which are symptomatic
* History of a decrease in LVEF to less than (<) 40% or symptomatic congestive heart failure (CHF) with previous trastuzumab treatment
* History of symptomatic CHF (New York Heart Association [NYHA] Classes II-IV) or serious cardiac arrhythmia requiring treatment
* History of myocardial infarction or unstable angina within 6 months of first study treatment
* Current dyspnea at rest due to complications of advanced malignancy or requirement for continuous oxygen therapy
* Current severe, uncontrolled systemic disease (clinically significant cardiovascular, pulmonary, or metabolic disease)
* Pregnancy or lactation
* Currently known active infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus
* History of intolerance (such as Grade 3-4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2185 (Actual)
Dates: Start 2012-11-27 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (300):
- Argentina (3):
  - CEMIC, Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Hospital Privado De Comunidad; General Practice, Mar del Plata
- Australia (8):
  - Mater Hospital; Patricia Ritchie Centre for Cancer Care and Research, North Sydney, New South Wales
  - Calvary Mater Newcastle; Medical Oncology, Waratah, New South Wales
  - Westmead Hospital; Medical Oncology and Pallative Care, Westmead, New South Wales
  - Haematology & Oncology Clinics of Australia Research Centre, South Brisbane, Queensland
  - Ashford Cancer Center Research, Kurralta Park, South Australia
  - Peter MacCallum Cancer Centre; Medical Oncology, Melbourne, Victoria
  - Sunshine Hospital; Oncology Research, St Albans, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (3):
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - Medizinische Universität Wien; Univ.Klinik für Frauenheilkunde - Klinik für Gynäkologie, Vienna
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I - Abt. für Onkologie, Vienna
- Belgium (10):
  - Institut Jules Bordet, Anderlecht
  - UZ Brussel, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - GHdC Site Notre Dame, Charleroi
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - CHU Sart-Tilman, Liège
  - Clinique Ste-Elisabeth, Namur
  - Sint Augustinus Wilrijk, Apotheek, Wilrijk
- Brazil (5):
  - *X*Instituto Nacional do Cancer - INCA, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Oncologicas - CEPON, Florianópolis, Santa Catarina
  - Hospital Sirio Libanes; Centro de Oncologia, São Paulo, São Paulo
  - Hospital Sao Jose, São Paulo, São Paulo
- Bulgaria (4):
  - MHAT Serdika; Department of medical oncology, Sofia
  - SHATO - Sofia, Sofia
  - SHATOD - Sofia, Sofia
  - District Oncology Dispensary Wit Stationary, Varna
- Canada (9):
  - BC Cancer - Surrey, Surrey, British Columbia
  - British Columbia Cancer Agency (Bcca) - Vancouver Cancer Centre, Vancouver, British Columbia
  - Dr. H. Bliss Murphy Cancer Centre; Oncology, St. John's, Newfoundland and Labrador
  - Royal Victoria Regional Health Centre; c/o Oncology Clinical Trials, Barrie, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Southlake Regional Health Center; Community Care Clinic / Oncology, Newmarket, Ontario
  - St. Michael'S Hospital, Toronto, Ontario
  - Hopital Maisonneuve- Rosemont; Oncology, Montreal, Quebec
  - Mcgill University - Royal Victoria Hospital; Oncology, Montreal, Quebec
- China (10):
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - Beijing Cancer Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Sun Yat-sen Memorial Hospital, Guangzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Cancer Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Zhejiang Cancer Hospital, Zhejiang
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- Denmark (7):
  - Aalborg Universitetshospital, Klinik Kirurgi-Kræft, Onkologisk afd., Aalborg
  - Herlev Hospital; Afdeling for Kræftbehandling, Herlev
  - Nordsjællands Hospital, Hillerød, Onkologisk Afdeling, Hillerød
  - Rigshospitalet; Onkologisk Klinik, København Ø
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense C
  - Sygehus Syd Roskilde; Onkologisk/haematologisk ambulatorium, Roskilde
  - Vejle Sygehus; Onkologisk Afdeling, Vejle
- Hospital Metropolitano de Santiago, Santiago de los Caballeros, Dominican Republic
- Ecuador (2):
  - Clinica Alcivar, torre 1;Private office, Guayaquil
  - Hospital Solca Portoviejo; Oncologia, Portoviejo
- North Estonia Medical Centre Foundation; Oncology Center, Tallinn, Estonia
- Finland (4):
  - Helsingin yliopistollinen keskussairaala, Helsinki
  - KYS Sadesairaala; Syopatautien poliklinikka, Kuopio
  - Tampere University Hospital; Dept of Oncology, Tampere
  - Turku Uni Central Hospital; Oncology Clinics, Turku
- France (40):
  - Clinique De L Europe; Radiotherapie Chimiotherapie, Amiens
  - ICO Paul Papin; Oncologie Medicale., Angers
  - Institut Sainte Catherine, Avignon
  - Hopital Jean Minjoz - CHU de Besançon, Besançon
  - Clinique Tivoli; Chimiotherapie Radiotherapie, Bordeaux
  - Institut Bergonie; Oncologie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine; Chimiotherapie Radiotherapie, Bordeaux
  - Cli De La Porte De Saint Cloud; Hop De Jour De Chimiotherapie, Boulogne-Billancourt
  - Hopital Morvan; Oncologie - Radiotherapie, Brest
  - Centre Francois Baclesse; Radiotherapie, Caen
  - Centre Jean Perrin; Oncologie, Clermont-Ferrand
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - Chu Grenoble - Hopital Albert Michallon; Departement de Cancero-Hematologie, Grenoble
  - Centre Hartmann, Levallois-Perret
  - Centre Oscar Lambret; Senologie, Lille
  - Clinique Chenieux; Oncology, Limoges
  - Ch Bretagne Sud Site Scorff; Oncologie Medicale, Lorient
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes; Oncologie Medicale, Marseille
  - Hopital Layne; Medecine Ambulatoire, Mont-de-Marsan
  - Centre Val Aurelle Paul Lamarque; Recherche Clinique, Montpellier
  - Centre Antoine Lacassagne; Hopital De Jour A2, Nice
  - Institut Curie; Oncologie Medicale, Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Centre Catalan D' Oncologie, Perpignan
  - Polyclinique Francheville; Med Chimiotherapie Radiotherapie, Périgueux
  - Clinique Armoricaine Radiologie; Hopital de Jour, Plérin
  - Pole Regional De Cancerologie, Poitiers
  - Institut Jean Godinot; Oncologie Medicale, Reims
  - Polyclinique De Courlancy; Centre Radiotherapie Oncologie, Reims
  - Centre Eugene Marquis; Unite Huguenin, Rennes
  - Centre Henri Becquerel; Oncologie Medicale, Rouen
  - Centre Rene Huguenin; CONSULT SPECIALISEES, Saint-Cloud
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Centre Paul Strauss; Oncologie Medicale, Strasbourg
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Clinique Pasteur; Oncologie Medicale, Toulouse
  - Centre Henry S Kaplan - CHU Bretonneau ; service oncologie, Tours
  - Centre Alexis Vautrin; Oncologie Medicale, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy; Pathologie Mammaire, Villejuif
- Germany (19):
  - Hämatologisch-onkologische Praxis Dr. med. - Heinrich, - Bangerter, Augsburg
  - Praxis Dres. Schilling & Till, Berlin
  - Schwerpunktpraxis Onkologie/Hämatologie Dr. Dirk Pott, Dr. Christian Tirier und Carla Verena u.w., Bottrop
  - Onkozentrum Dres. Göhler, Dresden
  - Dres. Joerg Weniger, Annette Bittrich und Berit Schuetze, Erfurt
  - Universitätsklinikum Erlangen; Frauenklinik, Erlangen
  - OncoResearch Lerchenfeld GmbH, Hamburg
  - HOPA MVZ GmbH, Hamburg
  - Medizinische Hochschule Zentrum Frauenheilkunde Abt.Gynäkologische Onkologie, Hanover
  - Institut für Versorgungsforschung in der Onkologie GbR Koblenz, Koblenz
  - Klinikum Leverkusen; Med. Klinik III / Onkologie, Leverkusen
  - Klinikum der Universität München; Campus Großhadern; Klinik und Poliklinik für Frauenheilkunde, München
  - Universitätsklinikum Münster; Klinik für Frauenheilkunde und Geburtshilfe, Münster
  - Sana Klinikum Offenbach GmbH; Klinik für Gynäkologie & Geburtshilfe, Offenbach
  - Praxis für Hämatologie und Onkologie, Porta Westfalica
  - Universitaetsfrauenklinik; Und Poliklinik Am Klinikum, Rostock
  - Universitätsklinik Tübingen; Frauenklinik, Tübingen
  - HELIOS Dr. Horst Schmidt Kliniken Wiesbaden; Klinik für Gynäkologie und gynäkologische Onkologie, Wiesbaden
  - Hämatologisch-Onkologische Schwerpunktpraxis Dres. Schlag & Schöttker, Würzburg
- Greece (4):
  - University General Hospital of Heraklion, Crete
  - Uni Hospital of Ioannina; Oncology Dept., Ioannina
  - University Hospital of Patras Medical Oncology, Pátrai
  - Papageorgiou General Hospital; Medical Oncology, Thessaloniki
- Centro Oncológico Sixtino / Centro Oncológico SA, Guatemala City, Guatemala
- Hong Kong (2):
  - Princess Margaret Hospital; Oncology, Hong Kong
  - Prince of Wales Hosp; Dept. Of Clinical Onc, Shatin
- Hungary (5):
  - Ogyi, Orszagos Gyogyszereszeti Intezet, Budapest
  - Szent Imre Hospital; Dept. of Oncology, Budapest
  - Orszagos Onkologiai Intezet; B Belgyogyaszati Osztaly, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont; Fázis I-es Klinikai Farmakológiai Vizsgálóhely, Budapest
  - Kaposi Mor County Hospital; Dept. of Oncology, Kaposvár
- Landspitali University Hospital, Department of Medical Oncology, Reykjavik, Iceland
- Indonesia (3):
  - Cipto Mangunkusumo General Hospital; Hematology & Oncology, Jakarta
  - Dharmais National Cancer Center, Jakarta
  - MRCCC Siloam Semanggi Hospital, Jakarta
- Ireland (4):
  - Cork Uni Hospital; Oncology Dept, Cork
  - St Vincent'S Uni Hospital; Medical Oncology, Dublin
  - Mater Misericordiae Uni Hospital; Oncology, Dublin
  - University Hospital Limerick - Oncology, Limerick
- Italy (31):
  - Ospedale Antonio Perrino; Oncologia Medica, Brindisi, Apulia
  - Ospedale Vito Fazzi; Div. Oncoematologia, Lecce, Apulia
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino, Campania
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Università degli Studi Federico II; Clinica di Oncologia Medica, Napoli, Campania
  - Ospedale Bellaria; U.O. Oncologia Medica, Bologna, Emilia-Romagna
  - A.O.U. Policlinico di Modena, Modena, Emilia-Romagna
  - Az. Osp. Ospedale Civile; U.O. Di Oncologia Medica Ed Ematologia, Piacenza, Emilia-Romagna
  - RCCS - Centro di Riferimento; Oncologia Medica B, Aviano (PN), Friuli Venezia Giulia
  - Divisione Onc Med dell'Azienda, Udine, Friuli Venezia Giulia
  - Policlinico Umberto i di Roma; dip. Scienze Radiologiche, Oncologiche, Anatomopatologiche, Rome, Lazio
  - Ospedale S.S. Trinità Nuovo; Divisione Oncologia, Sora, Lazio
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - ASST DI CREMONA; Unità di Patologia Mammaria Senologia e Breast Unit, Cremona, Lombardy
  - ASST DI LECCO; Oncologia Medica, Lecco, Lombardy
  - Ospedale San Raffaele; Medical Oncology, Milan, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 1, Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Fondazione Salvatore Maugeri; Divisione Di Oncologia Medica, Pavia, Lombardy
  - Casa di Cura Multimedica S.p.A.; Dipartimento Oncologico, Sesto San Giovanni (MI), Lombardy
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo; Dipartimento Oncologico, Candiolo, Piedmont
  - Ospedale Maggiore Della Carita; Oncologia Medica, Novara, Piedmont
  - A.O. Città della Salute e della Scienza - Presidio Molinette; divisione oncologia medica, Turin, Piedmont
  - Az Ospedaliera Nuovo Garibaldi Quartiere Nesima; Oncologia Medica, Catania, Sicily
  - A.O.U Careggi, Florence, Tuscany
  - Azienda usl 5 Di Pisa-Ospedale Di Pontedera;U.O. Oncologia, Pontedera, Tuscany
  - Ospedale Misericordia E Dolce; Oncologia Medica, Prato, Tuscany
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia; Oncologia Medica, Perugia, Umbria
  - Ospedale Civile; Oncologia Medica, Camposampiero, Veneto
  - Ospedale Busonera; Oncologia Medica, Padua, Veneto
  - A.O.U.I. VERONA-OSPEDALE BORGO TRENTO; ONCOLODIA MEDICA-d.O., Verona, Veneto
- CHL Hopital Municipal; Oncology, Luxembourg, Luxembourg
- Mexico (6):
  - Hospital General de México, Mexico City, Mexico CITY (federal District)
  - Medica Sur Centro Oncologico Integral, D.F.
  - Hospital Hmg Coyoacan, DF
  - CENTRO MÉDICO NACIONAL SIGLO XXI; Hospital de Especialidades Oncología, Mexico City
  - Inst. Nacional de Cancerologia; Investigacion Clinica, Mexico City
  - Instituto Nacional de Ciencias Médicas Y de La Nutricion Zubirán, Mexico City
- Netherlands (9):
  - Antoni Van Leeuwenhoek Ziekenhuis; Inwendige Geneeskunde, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Deventer Ziekenhuis; Interne Geneeskunde, Deventer
  - Ziekenhuisgroep Twente, Hengelo, Hengelo
  - Spaarne Ziekenhuis; Inwendige Geneeskunde, Hoofddorp
  - Medisch Centrum Leeuwarden; Interne, Leeuwarden
  - Orbis Medisch Centrum; Inwendige Geneeskunde, Sittard-Geleen
  - MC Haaglanden; Oncologie, The Hague
  - Twee Steden Ziekenhuis - Locatie Tilburg; Interne Geneesekunde, Tilburg
- Oslo Universitetssykehus HF; Ullevål sykehus, Oslo, Norway
- Panama (2):
  - Centro Hemato Oncologico Panama, Panama City
  - Centro Oncologico America, Panama City
- Peru (2):
  - Instituto;Oncologico Miraflores, Lima
  - Clinica de Especialidades Medicas, Lima
- Poland (6):
  - Bialostockie Centrum Onkologii; Oddzial Onkologii Klinicznej, Bialystok
  - Szpital Specjalistyczny POO im. ks. B.Markiewicza; Dzienny Oddz Chemioter i Hematologii Onkol, Brzozów
  - Świętokrzyskie Centrum Onkologii; Dział Chemioterapii, Kielce
  - Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Kliniki Onkologii, Krakow
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina, Klinika Onkologii, Otwock
  - Wojewódzki Szpital Specjalistyczny Nr 3, Rybnik
- Portugal (3):
  - IPO de Lisboa; Servico de Oncologia Medica, Lisbon
  - Hospital da Luz; Departamento de Oncologia Medica, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Slovakia (2):
  - Narodny Onkologicky Ustav; Oddelenie klinickej onkologie A, Bratislava
  - Fakultna nemocnica Trencín; Onkologicke odd., Trenčín
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Korea (5):
  - Kyungpook National University Medical Center, Daegu
  - Gachon Medical School Gil Medical Center; Medical Oncology, Incheon
  - Seoul National Uni Hospital; Dept. of Internal Medicine/Hematology/Oncology, Seoul
  - Yonsei University Severance Hospital; Medical Oncology, Seoul
  - Korea University Anam Hospital; Oncology Haemotology, Seoul
- Spain (33):
  - Hospital General Universitario de Elche; Servicio de Oncologia, Elche, Alicante
  - Hospital General de Elda; Servicio de Oncologia, Elda, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital de Jerez de la Frontera; Servicio de Oncologia, Jerez de la Frontera, Cadiz
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Hospital de Donostia; Servicio de Oncologia Medica, Donostia / San Sebastian, Guipuzcoa
  - Hospital Universitario Materno Infantil de Gran Canaria; Servicio de Oncologia, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital de Gran Canaria Dr. Negrin; Servicio de Oncologia, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Severo Ochoa; Servicio de Oncologia, Leganés, Madrid
  - Hospital Quiron de Madrid; Servicio de Oncologia, Pozuelo de Alarcón, Madrid
  - Hospital Xeral Cíes; Servicio de Oncologia, Vigo, Pontevedra
  - Hospital Univ. Central de Asturias; Servicio de Oncologia, Oviedo, Principality of Asturias
  - Hospital Universitari Sant Joan de Reus; Servicio de Oncologia, Reus, Tarragona
  - Hospital de Cruces; Servicio de Oncologia, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario A Coruña (CHUAC, Materno Infantil), Oncología, A Coruña
  - Hospital General Univ. de Alicante; Servicio de Oncologia, Alicante
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Quiron Barcelona; Servicio de Oncologia, Barcelona
  - Hospital San Pedro De Alcantara; Servicio de Oncologia, Cáceres
  - Hospital Universitari de Girona Dr. Josep Trueta; Servicio de Oncologia, Girona
  - Hospital Universitario San Cecilio; Servicio de Oncologia, Granada
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Hospital Universitari Arnau de Vilanova de Lleida; Servicio de Oncologia, Lleida
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Complejo Hospitalario de Pontevedra; Servicio de Oncologia, Pontevedra
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
  - Hospital General Universitario de Valencia; Servicio de oncologia, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Sweden (2):
  - Karolinska Hospital; Oncology - Radiumhemmet, Stockholm
  - Norrlands universitetssjukhus; Onkologkliniken, Umeå
- Taiwan (3):
  - National Cheng Kung Uni Hospital; Surgery, Tainan
  - Chi-Mei Medical Centre; Hematology & Oncology, Tainan
  - VETERANS GENERAL HOSPITAL; Department of General Surgery, Taipei
- Thailand (3):
  - Department of Surgery, King Chulalongkorn Memorial Hospital, Bangkok
  - Pramongkutklao Hospital; Medicine - Medical Oncology Unit, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital; Department of Surgery/Head Neck and Breast Unit; Clinical Trial, Chiang Mai
- Turkey (Türkiye) (10):
  - Gazi Uni Medical Faculty Hospital; Oncology Dept, Ankara
  - Gaziantep University Medical Faculty, Medical Oncology Department, Gaziantep
  - Bezmialem Vakif Univ Medical; Bezmialem Vakif Univ T, Istanbul
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital; Medical Oncology, Istanbul
  - Istanbul Uni of Medicine Faculty; Oncology Dept, Istanbul
  - Kartal Dr Lutfi Kirdar Sehir Hastanesi; Medical Oncology Department, Istanbul
  - Marmara Uni Faculty of Medicine; Medical Oncology, Istanbul
  - Ege Uni Medical Faculty Hospital; Oncology Dept, Izmir
  - Dokuz Eylul Uni ; Medical Oncology, Izmir
  - Kocaeli University Faculty of Medicine; Medical oncology, İzmit
- Tawam Hospital, Al Ain City, United Arab Emirates
- United Kingdom (29):
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospital Birmingham Queen Elizabeth Hospital, Birmingham
  - Kent & Canterbury Hospital, Canterbury
  - University Hospital coventry; Oncology Department, Coventry
  - Eastborne District General Hospital, Eastbourne
  - Western General Hospital; Clinical Oncology, Edinburgh
  - St Margaret'S Hospital; Breast Unit, Epping
  - Royal Devon & Exeter Hospital; Oncology Centre, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Diana Princess of Wales Hosp., Grimsby
  - Huddersfield Royal Infirmary, Huddersfield
  - Castle Hill Hospital; The Queen's Centre for Oncology & Haematology, Hull
  - Ipswich Hospital; Oncology Pharmacy, Ipswich
  - Royal Lancaster Infirmary, Morecambe Bay Hospitals Nhs Trust, Lancaster
  - Royal Free Hospital; Dept of Oncology, London
  - Guys & St Thomas Hospital; Department of Oncology, London
  - St George'S Hospital; Oncology Research Office /Oncology Opd, London
  - Sarah Cannon Research Institute, London
  - Maidstone & Tonbridge Wells Hospital; Kent Oncology Center, Maidstone
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - Mount Vernon Hospital, Middlesex
  - Plymouth Oncology Centre; Clinical Trials Unit, Plymouth
  - Queen Alexandra Hospital, Portsmouth, Portsmouth
  - Queen's Hospital; Oncology, Romford
  - Weston Park Hospital; Cancer Clinical Trials Centre, Sheffield
  - Royal Shrewsbury Hospital, Shrewsbury
  - Singleton Hospital; Pharmacy, Swansea
  - Yeovil District Hospital; Macmillan Cancer Unit, Yeovil
  - York District Hospital, York
- Venezuela (3):
  - Unidad de Mastologia y Atencion a la Mujer, Barcelona
  - Instituto Oncológico Luis Razetti, Caracas
  - Instituto de Oncologia y Hematologia UCV, Caracas

REFERENCES:
- [Derived] Wuerstlein R, Ellis P, Montemurro F, Anton Torres A, Delaloge S, Zhang Q, Wang X, Wang S, Shao Z, Li H, Rachman A, Vongsaisuwon M, Liu H, Fear S, Pena-Murillo C, Barrios C. Final results of the global and Asia cohorts of KAMILLA, a phase IIIB safety trial of trastuzumab emtansine in patients with HER2-positive advanced breast cancer. ESMO Open. 2022 Oct;7(5):100561. doi: 10.1016/j.esmoop.2022.100561. Epub 2022 Sep 7. PMID 36084395
- [Derived] Engebraaten O, Yau C, Berg K, Borgen E, Garred O, Berstad MEB, Fremstedal ASV, DeMichele A, Veer LV', Esserman L, Weyergang A. RAB5A expression is a predictive biomarker for trastuzumab emtansine in breast cancer. Nat Commun. 2021 Nov 5;12(1):6427. doi: 10.1038/s41467-021-26018-z. PMID 34741021
- [Derived] Montemurro F, Delaloge S, Barrios CH, Wuerstlein R, Anton A, Brain E, Hatschek T, Kelly CM, Pena-Murillo C, Yilmaz M, Donica M, Ellis P. Trastuzumab emtansine (T-DM1) in patients with HER2-positive metastatic breast cancer and brain metastases: exploratory final analysis of cohort 1 from KAMILLA, a single-arm phase IIIb clinical trial☆. Ann Oncol. 2020 Oct;31(10):1350-1358. doi: 10.1016/j.annonc.2020.06.020. Epub 2020 Jul 5. PMID 32634611

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort 1 has 2003 participants and Cohort 2 has 182 participants representing the total enrollment study number. Cohort 1 was conducted in 281 centers in 40 countries worldwide whereas Cohort 2 was conducted in an Asian population in 14 centers in China, Thailand and Indonesia.
Pre-assignment Details: Two participants (one in Corhort 1 and Corhot 2) were not included in the safety population as one didn't receive study treatment and one did not qualify under the inclusion criteria.
Groups:
- Trastuzumab Emtansine (All Participants): This cohort (Cohort 1) enrolled all participants with HER2 positive, unresectable, LABC or mBC who had received prior anti-HER2 and chemotherapy treatment and had progressed on or after the most recent treatment for LABC or mBC, or within 6 months of completing adjuvant therapy. Participants received trastuzumab emtansine every 3 weeks until unacceptable toxicity, withdrawal of consent, or disease progression.
- Trastuzumab Emtansine (Asian Participants): This cohort (Cohort 2) enrolled Asian race participants with HER2-positive, unresectable, LABC or mBC who had received prior anti-HER2 and chemotherapy treatment and had progressed on or after the most recent treatment for LABC or mBC, or within 6 months of completing adjuvant therapy. Participants received trastuzumab emtansine every 3 weeks until unacceptable toxicity, withdrawal of consent, or disease progression.
Period: Overall Study
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants)
Started | 2003 | 182
Completed | 494 (For one participant, the site incorrectly answered the question 'Did the participant complete follow-up as per protocol?' It was answered No, however the participant was in survival follow-up and the site should have answered Yes. This participant is wrongly counted in the 'discontinued from study' number.) | 65
Not Completed | 1509 | 117
Not completed — Death | 1067 | 76
Not completed — Lost to Follow-up | 144 | 10
Not completed — Adverse Event/Unacceptable Toxicity | 4 | 0
Not completed — Investigator Decision | 5 | 0
Not completed — Not Classifiable | 1 | 0
Not completed — On Study Treatment At Lplv/Cohort 1 | 93 | 0
Not completed — On Study Treatment At Lplv/Cohort 2 | 0 | 1
Not completed — Progressive Disease | 3 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Safety FU Done < 3 Months Prior To CCOD | 9 | 1
Not completed — Termination By Sponsor | 4 | 0
Not completed — Withdrawal by Subject | 177 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants) | Total
Number analyzed (Participants) | 2003 | 182 | 2185
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (11.4) | 49.1 (10.1) | 54.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1989 | 182 | 2171
  Male | 14 | 0 | 14
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    Caucasian | 1397 | 0 | 1397
    Black | 21 | 0 | 21
    Asian | 72 | 182 | 254
    Native American | 41 | 0 | 41
    N/A as per local regulation | 466 | 0 | 466
    Unknown | 3 | 0 | 3
    Other | 2 | 0 | 2
    Missing | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity
  Participants
    Hispanic/Latino | 300 | 0 | 300
    Chinese | 29 | 147 | 176
    N/A as per local regulation | 997 | 16 | 1013
    Other | 417 | 19 | 436
    Mixed | 9 | 0 | 9
    Indian (Indian subcontinent) | 4 | 0 | 4
    Unknown | 247 | 0 | 247

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events of Primary Interest (AEPIs)
Description: The AEPIs in this study were defined as the following: adverse events (AEs) Grade >/= 3, specifically, hepatic events, allergic reactions, thrombocytopenia and hemorrhage events, all Grade >/= 3 AEs related to trastuzumab emtansine and pneumonitis events of all grades.
Time Frame: Baseline up to approximately 7 years
Population: The safety population included all participants who had received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants)
Number analyzed (Participants) | 2002 | 181
Percentage of Participants | 23.1 [21.2 to 25.0] | 51.4 [43.9 to 58.9]

2. Secondary Outcome: Percentage of Participants With Specific AEPIs
Description: as for outcome 1
Time Frame: Baseline up to approximately 7 years
Population: The safety population included all participants who had received at least 1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants)
Number analyzed (Participants) | 2002 | 181
Percentage of Participants
  AEs Grade >/= 3 for hepatic events | 6.9 | 12.2
  AEs Grade >/= 3 for allergic reactions | 2.3 | 1.1
  AEs Grade >/= 3 for thrombocytopenia | 3.7 | 36.5
  AEs Grade >/= 3 for hemorrhage events | 2.3 | 1.7
  AEs Grade >/= 3 related to trastuzumab emtansine | 18.4 | 48.6
  Pneumonitis of all grades | 1.0 | 2.2

3. Secondary Outcome: Percentage of Participants With Adverse Events of Special Interest (AESIs)
Description: AESIs included: 1) Potential drug-induced liver injury, which included any potential case of drug-induced liver injury as, assessed by laboratory criteria for Hy's law (AST and/or ALT elevations that were >3 × ULN, Concurrent elevation of total bilirubin >2 × ULN (or clinical jaundice if total bilirubin measures were not available), except in participants with documented Gilbert's syndrome. Those with Gilbert's syndrome, elevation of direct bilirubin >2 × ULN was used instead. 2) Suspected transmission of an infectious agent by study drug was defined as any organism, virus, or infectious particle (e.g., prion protein transmitting transmissible spongiform encephalopathy), pathogenic or non-pathogenic. A transmission of an infectious agent suspected from clinical symptoms or laboratory findings indicating an infection in a participant exposed to a medicinal product.
Time Frame: Baseline up to approximately 7 years
Population: The safety population included all participants who had received at least 1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants)
Number analyzed (Participants) | 2002 | 181
Percentage of Participants
  Potential drug-induced liver injury | 1.2 | 1.1
  Suspected transmission of an infectious agent | 0.2 | 0.0

4. Secondary Outcome: Progression-Free Survival According to Response Evaluation for Solid Tumors (RECIST) Version (v) 1.1 As Per Investigator Assessment
Description: Progression free survival is defined as the time (in months) between the date of first dose and the date of disease progression or death from any cause. Progressive disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm).
Time Frame: Baseline up to disease progression or death due to any cause, whichever occurs first (assessed every 12 weeks during treatment period thereafter 28-42 days after the last dose or every 3-6 months up to approximately 7 years)
Population: Intent to Treat (ITT) Population included all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants)
Number analyzed (Participants) | 2003 | 182
months | 6.8 [5.8 to 7.6] | 5.7 [5.5 to 7.0]

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time to death, which is the time from the date of dosing until the date of death, regardless of the cause of death.
Time Frame: Baseline until death (up to approximately 7 years)
Population: ITT Population included all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants)
Number analyzed (Participants) | 2003 | 182
months | 27.2 [25.5 to 28.7] | 29.5 [21.1 to NA] — The confidence interval has no upper limit

6. Secondary Outcome: Percentage of Participants With Best Overall Response (Complete Response [CR] or Partial Response [PR]) According to RECIST v 1.1 As Per Investigator Assessment
Description: Best Overall Response reported here is the Best confirmed Overall Response. To be assigned a status of PR or CR, i.e., to be a responder, changes in tumor measurements had to be confirmed by repeat assessments that had to be performed no less than 4 weeks after the criteria for response were first met, i.e., participants needed to have two consecutive assessments of PR or CR. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: as for outcome 4
Population: ITT Population included all participants enrolled in the study. Only participants with measurable disease were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants)
Number analyzed (Participants) | 1613 | 169
Percentage of Participants | 29.3 [27.1 to 31.6] | 29.6 [22.8 to 37.1]

7. Secondary Outcome: Percentage of Participants With Clinical Benefit (CR or PR or Stable Disease [SD]) According to RECIST v 1.1
Description: Clinical Benefit was defined as CR plus PR plus SD. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. SD: neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants)
Number analyzed (Participants) | 1613 | 169
Percentage of Participants | 47.1 [44.7 to 49.6] | 39.6 [32.2 to 47.4]

8. Secondary Outcome: Duration of Response (DOR) According to RECIST v 1.1
Description: DOR is defined as the period from the date of initial confirmed PR or CR (whichever occurs first) until the date of PD or death from any cause. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm).
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants)
Number analyzed (Participants) | 1613 | 169
months | 13.8 [12.2 to 15.0] | 14.2 [11.1 to 24.4]

9. Secondary Outcome: Time to Response According to RECIST v 1.1
Description: Time to Response is defined as the time from first dose to first documentation of confirmed PR or CR (whichever occurs first). CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: as for outcome 4
Population: ITT Population included all participants enrolled in the study. Only responders were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants)
Number analyzed (Participants) | 473 | 50
months | 22.3 [11.8 to 38.2] | 8.3 [5.7 to NA] — The confidence interval has no upper limit

10. Secondary Outcome: Number of Hospital Visits
Description: The number of hospital visits were recorded to evaluate the resoruce expenditures while participants were on study treatment.
Time Frame: Baseline up to approximately 7 years
Population: The safety population included all participants who had received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Number of Hospital Visits
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants)
Number analyzed (Participants) | 2002 | 181
Number of Hospital Visits | 2.7 (2.78) | 2.1 (1.70)

11. Secondary Outcome: Type of Hospital Visits
Description: The type of hospital visits (intensive care unit (ICU) versus other) were recorded to evaluate the resoruce expenditures while participants were on study treatment. The number of participants with at least one ICU visit are based on the number of participants with at least one hospital visit, in each group.
Time Frame: Baseline up to approximately 7 years
Population: The safety population included all participants who had received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants)
Number analyzed (Participants) | 2002 | 181
Participants
  Other Hospital Visit | 558 | 33
  ICU Visit: number analyzed (Participants) | 558 | 33
  ICU Visit | 39 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 7 years
Description: The analysis of AEs focused on treatment-emergent AEs (TEAEs) which were AEs that occurred on the day of or after first administration of study drug.
Arm/Group | Trastuzumab Emtansine (All Participants) | Trastuzumab Emtansine (Asian Participants)
All-Cause Mortality (participants affected / at risk) | 1072/2002 | 77/181
Serious Adverse Events (participants affected / at risk) | 427/2002 | 36/181
Other Adverse Events (participants affected / at risk) | 1734/2002 | 170/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab Emtansine (All Participants) (N=2002) | Trastuzumab Emtansine (Asian Participants) (N=181)
ANAEMIA (Blood and lymphatic system disorders) | 13 (14) | 0 (0)
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 11 (11) | 10 (11)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 3 (3) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC TAMPONADE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 1 (1) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 2 (2) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 (2) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 3 (3) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
BLINDNESS (Eye disorders) | 1 (2) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 1 (1)
RETINAL VEIN THROMBOSIS (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (12) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 0 (0)
ANAL FISSURE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (4) | 0 (0)
ASCITES (Gastrointestinal disorders) | 2 (6) | 0 (0)
COLITIS (Gastrointestinal disorders) | 3 (3) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 3 (3) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 2 (2) | 0 (0)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (2) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 2 (3) | 0 (0)
GASTRIC ANTRAL VASCULAR ECTASIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1 (10) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 3 (3) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRODUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (10) | 0 (0)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0)
GLOSSITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (3) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (2) | 1 (2)
MELAENA (Gastrointestinal disorders) | 2 (8) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 5 (6) | 1 (1)
OESOPHAGEAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 (4) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (3) | 0 (0)
PERIODONTAL DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (2) | 0 (0)
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (2) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
SUBILEUS (Gastrointestinal disorders) | 2 (4) | 0 (0)
TOOTH LOSS (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (6) | 2 (6)
VOMITING (Gastrointestinal disorders) | 17 (19) | 1 (1)
ASTHENIA (General disorders) | 3 (3) | 0 (0)
CATHETER SITE ERYTHEMA (General disorders) | 1 (1) | 0 (0)
CHILLS (General disorders) | 2 (6) | 0 (0)
DEATH (General disorders) | 5 (5) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 4 (4) | 0 (0)
HYPERTHERMIA (General disorders) | 2 (2) | 0 (0)
IMPLANT SITE DEHISCENCE (General disorders) | 1 (1) | 0 (0)
INFLAMMATION (General disorders) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 3 (3) | 1 (1)
PYREXIA (General disorders) | 13 (42) | 0 (0)
SUDDEN DEATH (General disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 3 (3) | 0 (0)
CHOLESTASIS (Hepatobiliary disorders) | 2 (2) | 0 (0)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 (3) | 1 (3)
HEPATIC FAILURE (Hepatobiliary disorders) | 5 (10) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC PAIN (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATOTOXICITY (Hepatobiliary disorders) | 7 (14) | 0 (0)
JAUNDICE (Hepatobiliary disorders) | 1 (1) | 0 (0)
NODULAR REGENERATIVE HYPERPLASIA (Hepatobiliary disorders) | 3 (6) | 0 (0)
NON-CIRRHOTIC PORTAL HYPERTENSION (Hepatobiliary disorders) | 1 (2) | 0 (0)
PORTAL HYPERTENSION (Hepatobiliary disorders) | 2 (4) | 0 (0)
ALLERGIC OEDEMA (Immune system disorders) | 1 (3) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 2 (6) | 0 (0)
ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ACINETOBACTER INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ARTHRITIS INFECTIVE (Infections and infestations) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
BACTERIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
BACTERIAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
BRAIN ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
BREAST CELLULITIS (Infections and infestations) | 2 (2) | 0 (0)
BRONCHITIS (Infections and infestations) | 3 (4) | 0 (0)
CATHETER SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 8 (10) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 1 (1) | 0 (0)
DENGUE HAEMORRHAGIC FEVER (Infections and infestations) | 0 (0) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 6 (6) | 0 (0)
ENCEPHALITIS (Infections and infestations) | 1 (1) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 2 (2) | 0 (0)
ERYSIPELAS (Infections and infestations) | 4 (5) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 0 (0)
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 2 (2) | 0 (0)
INFECTION (Infections and infestations) | 3 (3) | 0 (0)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 1 (1) | 0 (0)
INFECTIVE EXACERBATION OF BRONCHIECTASIS (Infections and infestations) | 1 (1) | 0 (0)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1 (1) | 0 (0)
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
LISTERIOSIS (Infections and infestations) | 1 (1) | 0 (0)
LIVER ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (10) | 0 (0)
MASTITIS (Infections and infestations) | 2 (2) | 0 (0)
MENINGITIS (Infections and infestations) | 1 (1) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 3 (3) | 0 (0)
PERITONITIS (Infections and infestations) | 2 (2) | 0 (0)
PHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1)
PNEUMOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 22 (23) | 8 (8)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 2 (2) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 (1) | 0 (0)
PYELONEPHRITIS CHRONIC (Infections and infestations) | 1 (2) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 9 (9) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 2 (2) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 2 (2) | 0 (0)
STREPTOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
TRACHEOBRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (4) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 11 (12) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 3 (3) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (2) | 0 (0)
VULVAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ANASTOMOTIC ULCER (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 8 (8) | 0 (0)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 2 (6) | 0 (0)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RADIATION NECROSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SKELETAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPLENIC INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 0 (0)
AMYLASE INCREASED (Investigations) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (4) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 2 (2) | 1 (1)
ECG SIGNS OF MYOCARDIAL ISCHAEMIA (Investigations) | 1 (1) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 3 (3) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 3 (3) | 0 (0)
LIVER FUNCTION TEST INCREASED (Investigations) | 0 (0) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 2 (2) | 8 (12)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BONE LESION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
HAEMATOMA MUSCLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
KYPHOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BENIGN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTATIC UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NAEVUS HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SKIN NEOPLASM BLEEDING (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
APHASIA (Nervous system disorders) | 2 (4) | 0 (0)
ATAXIA (Nervous system disorders) | 1 (1) | 0 (0)
BRAIN OEDEMA (Nervous system disorders) | 6 (7) | 0 (0)
CENTRAL NERVOUS SYSTEM NECROSIS (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 4 (8) | 1 (2)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 2 (2) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (2) | 0 (0)
DIZZINESS (Nervous system disorders) | 3 (4) | 0 (0)
EPILEPSY (Nervous system disorders) | 8 (15) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 3 (6) | 0 (0)
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 (2) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 5 (5) | 0 (0)
IIIRD NERVE PARESIS (Nervous system disorders) | 1 (1) | 0 (0)
LEUKOENCEPHALOPATHY (Nervous system disorders) | 2 (2) | 0 (0)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0)
MOTOR DYSFUNCTION (Nervous system disorders) | 1 (1) | 0 (0)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
PARTIAL SEIZURES (Nervous system disorders) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 2 (2) | 0 (0)
SCIATICA (Nervous system disorders) | 2 (2) | 0 (0)
SEIZURE (Nervous system disorders) | 7 (11) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0)
VOCAL CORD PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
DEVICE BREAKAGE (Product Issues) | 1 (1) | 0 (0)
DEVICE EXTRUSION (Product Issues) | 1 (1) | 0 (0)
DEVICE LOOSENING (Product Issues) | 1 (1) | 0 (0)
AGITATION (Psychiatric disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 2 (2) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 4 (4) | 0 (0)
DEPRESSION (Psychiatric disorders) | 3 (4) | 0 (0)
HALLUCINATION (Psychiatric disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 2 (4) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 2 (2) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 4 (4) | 0 (0)
RENAL INJURY (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
CYSTOCELE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
METRORRHAGIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
UTERINE POLYP (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 1 (1)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHOKING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 (24) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
PULMONARY ALVEOLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RESPIRATORY TRACT HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SPIDER NAEVUS (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
BREAST CONSERVING SURGERY (Surgical and medical procedures) | 1 (1) | 0 (0)
SCAR EXCISION (Surgical and medical procedures) | 1 (1) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (3) | 0 (0)
EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 2 (2) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (3) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
VENA CAVA THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab Emtansine (All Participants) (N=2002) | Trastuzumab Emtansine (Asian Participants) (N=181)
ANAEMIA (Blood and lymphatic system disorders) | 173 (231) | 27 (49)
LEUKOPENIA (Blood and lymphatic system disorders) | 19 (23) | 15 (69)
NEUTROPENIA (Blood and lymphatic system disorders) | 79 (151) | 17 (72)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 165 (257) | 47 (157)
ABDOMINAL PAIN (Gastrointestinal disorders) | 139 (182) | 6 (8)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 135 (163) | 5 (5)
CONSTIPATION (Gastrointestinal disorders) | 394 (568) | 10 (38)
DIARRHOEA (Gastrointestinal disorders) | 252 (376) | 9 (9)
DRY MOUTH (Gastrointestinal disorders) | 283 (303) | 7 (13)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 83 (96) | 14 (19)
NAUSEA (Gastrointestinal disorders) | 651 (1204) | 28 (45)
STOMATITIS (Gastrointestinal disorders) | 160 (213) | 4 (6)
VOMITING (Gastrointestinal disorders) | 294 (408) | 17 (24)
ASTHENIA (General disorders) | 491 (828) | 18 (44)
FATIGUE (General disorders) | 556 (846) | 12 (17)
INFLUENZA LIKE ILLNESS (General disorders) | 107 (161) | 3 (3)
OEDEMA PERIPHERAL (General disorders) | 102 (115) | 6 (10)
PAIN (General disorders) | 85 (92) | 10 (11)
PYREXIA (General disorders) | 339 (1599) | 47 (243)
NASOPHARYNGITIS (Infections and infestations) | 136 (195) | 8 (13)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 80 (107) | 14 (18)
URINARY TRACT INFECTION (Infections and infestations) | 157 (230) | 4 (4)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 86 (100) | 58 (133)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 136 (156) | 77 (143)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 52 (52) | 14 (16)
BLOOD BILIRUBIN INCREASED (Investigations) | 89 (171) | 30 (85)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 84 (94) | 21 (31)
NEUTROPHIL COUNT DECREASED (Investigations) | 36 (58) | 20 (84)
PLATELET COUNT DECREASED (Investigations) | 91 (124) | 55 (191)
TRANSAMINASES INCREASED (Investigations) | 27 (28) | 18 (39)
WEIGHT DECREASED (Investigations) | 106 (109) | 8 (8)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 11 (13) | 20 (85)
DECREASED APPETITE (Metabolism and nutrition disorders) | 320 (398) | 16 (23)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 13 (13) | 11 (14)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 73 (91) | 19 (37)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 265 (349) | 6 (7)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 199 (226) | 5 (5)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 124 (154) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 135 (150) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 205 (279) | 8 (11)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 148 (169) | 3 (3)
DIZZINESS (Nervous system disorders) | 117 (137) | 11 (17)
HEADACHE (Nervous system disorders) | 454 (650) | 19 (32)
PARAESTHESIA (Nervous system disorders) | 128 (139) | 4 (5)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 113 (132) | 0 (0)
INSOMNIA (Psychiatric disorders) | 118 (134) | 11 (13)
COUGH (Respiratory, thoracic and mediastinal disorders) | 220 (256) | 23 (28)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 211 (705) | 2 (6)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 402 (669) | 30 (43)
HYPERTENSION (Vascular disorders) | 96 (113) | 12 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT01702571/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT01702571/SAP_001.pdf